CLINICAL TRIAL: NCT03218124
Title: Optimal Effect Site Remifentanil Concentration for Smooth Extubation After Thyroid Surgery
Brief Title: Optimal Remifentanil Concentration and Thyroidectomy
Acronym: ORCO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Prof. Gabriele Finco, Professor of Anesthesiology and Intensive Care, University of Cagliari
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Remismooth2217
Record Dates: First submitted 2017-07-10; First posted 2017-07-14 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Anesthesia
Keywords: Thyroidectomy; Remifentanil; Extubation; Cough; Target controlled infusion
MeSH Terms: conditions — Cough

STUDY DESIGN:
Intervention Model Description: Prospective observational study. Decreasing/increasing remifentanil effect site concentrations (Dixon's up and down model) to obtain cough-free extubation after thyroidectomy
Masking Description: Patient under general anesthesia unaware of the effect site concentration of remifentanil before extubation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- remifentanil (Experimental): After skin suture, a predetermined Effect site remifentanil concentration will be achieved. Starting from 1.5 ng/ml in the first patient and increased or decreased by 0.2 ng/ml intervals based on the previous patient response: up if cough present, down otherwise ("Dixon's up and down" method).
  Interventions: Other: Remifentanil Effect site concentration

INTERVENTIONS:
Other: Remifentanil Effect site concentration — After skin suture, a predetermined Effect site remifentanil concentration will be achieved. Starting from 1.5 ng/ml in the first patient and increased or decreased by 0.2 ng/ml intervals based on the previous patient response: up if cough present, down otherwise ("Dixon's up and down" method).

SUMMARY:
The study is aimed at determining the remifentanil effect site concentration suppressing the cough at extubation after surgical thyroidectomy, performed under remifentanil/desflurane based general anesthesia, expressed as median and 95th percentile effective dose.

Possible hemodynamic instability, respiratory depression or prolongation of awakening time are also sought.

ELIGIBILITY:
Inclusion Criteria:

* 18<age<67
* 6 hrs fasting
* American society of anesthesiology (ASA) Physical Status I o II
* Informed consent

Exclusion Criteria:

* Absence of inclusion criteria
* Use of cough suppressors, angiotensin converting enzyme-inhibitors, sedatives 4 weeks before surgery
* Arhythmia, pacemaker or unstable cardiovascular disease
* Hepatic or renal failure
* Anticipated difficulty in airways management
* Chronic obstructive pulmonary disease (COPD), Asthma, increased risk for inhalation, airway infection in the previous 4 weeks;
* Smoker
* Obesity (BMI >35)
* Pregnancy
* Hypersensitivity to drugs administered for the study

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-07-01 (Estimated)

PRIMARY OUTCOMES:
Cough | 15 minutes after surgery
  Any episode of sudden and violent abdominal contraction interrupting normal quite spontaneous or assisted ventilation would be accounted as "cough" and defines non-smooth extubation

SECONDARY OUTCOMES:
Hemodynamics 1 | 15 minutes after surgery
  Heart Rate (bpm)
Hemodynamics 2 | 15 minutes after surgery
  Blood pressure (mmHg)
Respiratory outcome 1 | 15 minutes after surgery
  Tidal Volume (ml)
Respiratory outcome 2 | 15 minutes after surgery
  End Tidal Carbon Dioxide (mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Finco, MD, Principal Investigator — Cagliari University
Locations (1):
- Policlinico Duilio Casula, Monserrato, Cagliari, Italy

IPD SHARING:
Plan to Share IPD: Undecided